CLINICAL TRIAL: NCT05390528
Title: A Phase I/II Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics and Initial Efficacy of HLX301(TIGIT×PDL1 Bispecific) in Patients With Locally Advanced/Metastatic Solid Tumors or Lymphoma
Brief Title: A Study Evaluating the Safety, Tolerability, Pharmacokinetic and Efficacy of HLX301(TIGIT×PDL1 Bispecific) in Locally Advanced/Metastatic Solid Tumors or Lymphoma
Acronym: HLX301
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX301-002
Record Dates: First submitted 2022-04-25; First posted 2022-05-25 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-04

CONDITIONS: Advanced Tumors; Lymphoma; Metastatic Tumors
MeSH Terms: conditions — Lymphoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group(phase Ia) (Experimental): Phase 1a uses accelerated titration design and Bayesian optimal interval (BOIN) design to investigate the safety of HLX301 and determine MTD.Six dose levels of 0.25 mg/kg, 1 mg/kg, 2.5 mg/kg, 5 mg/kg, 10 mg/kg, and 20mg/kg are planned for dose finding.
  Interventions: Drug: HLX301

INTERVENTIONS:
Drug: HLX301 — HLX301 will be administered as a single intravenous (IV) infusion on Day1 in each 14-day cycle.
  Other Names: A Recombinant Humanized Anti-PDL1 and Anti-TIGIT Bispecific Antibody

SUMMARY:
A Phase 1/2 Study of HLX301, A Recombinant Humanized Anti-PDL1 and Anti-TIGIT Bispecific Antibody, in patients with locally advanced/metastatic solid tumors or lymphoma.Up to 150 patients will be included in this study. Up to 30 DLT evaluable patients will be enrolled in phase 1a (dose escalation), 40 per-protocol treated patients in phase 1b (dose expansion), and 80 per-protocol treated patients in phase 2. Phase 1a to evaluate safety, dose limiting toxicity (DLT), and the maximum tolerated dose (MTD) of HLX301 in patients with advanced or metastatic tumors who have failed or are intolerant to standard therapy, or for whom no standard therapy is available.Phase 1b to identify the recommended phase 2 dose (RP2D) of HLX301 in patients with advanced or metastatic NSCLC who have failed or are intolerant to standard therapy, or for whom no standard therapy is available.

Phase 2 to evaluate the anti-tumor activity of HLX301 in patients with histologically or cytologically-confirmed non-small cell lung cancer (NSCLC), gastric/esophagogastric junction adenocarcinoma (GC/EGJ), head and neck squamous cell carcinoma (HNSCC), or urothelial carcinoma (UC) tumors that express PD-L1, after one or two prior systemic treatments and without standard therapy。

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet each of the following criteria are eligible for inclusion:

1. Patients who meet the following criteria will be enrolled:

   Phase 1a dose escalation: patients must have histologically or cytologically confirmed malignant solid tumors which are advanced or metastatic, have failed prior standard treatment, and be intolerant or ineligible for standard therapy (with the exception of hepatocellular carcinoma, which meets diagnostic criteria by dynamic CT/MRI).
2. Age ≥ 18 years, or legally an adult as per local regulations.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Measurable disease according to RECIST Version 1.1
5. Able to provide informed consent.
6. A life expectancy longer than three months.
7. Adequate hematologic parameters, defined as white blood cell count ≥ 3000/mm3 and absolute neutrophil counts ≥ 1500/mm3; hemoglobin≥9gm/dL; platelet count ≥ 90,000/mm3 without platelet transfusion within 14 days.
8. Adequate hepatic function, defined as serum albumin ≥ 3.0 g/dL; serum total bilirubin ≤ 1.5x upper limit of normal (ULN); serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN (AST and ALT ≤ 5 × ULN for patients with known liver metastasis or primary hepatocellular carcinoma); Child-Pugh score A in HCC.
9. Adequate renal function, defined as serum creatinine ≤ 1.5x upper limit of normal (ULN).
10. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 50% measured by cardiac ultrasound or MUGA scan; normal ECG or ECG without any clinically significant findings.

Exclusion Criteria:

* Exclusion criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Received prior anti-TIGIT therapy.
2. Patients who still have persistent ≥ grade 2 toxicities from prior therapies.
3. Concurrent unstable or uncontrolled medical conditions including, but not limited to, the following:

   i. Ongoing or active systemic infections requiring antibiotic treatment ii. Clinically significant arrhythmia, unstable angina pectoris, class III or IV congestive heart failure as per the New York Heart Association, or acute myocardial infarction in the past 6 months iii. Unhealed wound or ulcers persisting ≥ 3 months iv. Psychiatric illness or a social situation that would preclude study compliance v. Any other diseases, metabolic dysfunction, physical examination findings, or laboratory results raising reasonable suspicion of a disease or condition that contraindicates use of the investigational drug, that may affect interpretation of results, or that may place the patient at high risk of treatment complications.
4. Active CNS metastasis indicated by clinical symptoms, cerebral edema, steroid requirements (not including maintenance low dose steroids), or progressive growth.
5. History of any secondary malignancy in the past 2 years with the exception of curatively treated non-melanoma skin cancer or treated cervical carcinoma in situ.
6. Active or a history of (in the past 2 years) of autoimmune disease or syndrome requiring systemic steroid or immunosuppressive agents.
7. History of interstitial lung disease.
8. Hepatitis B virus infection (HBsAg or anti-HBc positive, and HBV-DNA positive), hepatitis C virus infection (anti-HCV positive, and HCV-RNA positive), or co-infection with hepatitis B and hepatitis C (positive HBsAg or anti-HBc, and positive anti-HCV).
9. Human immunodeficiency virus (HIV) infection.
10. Major surgery, treatment with anti-cancer or investigational agents, or radiotherapy in the 28 days prior to the first study dosing.
11. Treatment with immune check point inhibitors (anti-PD-1 or anti-PD-L1) in the 42 days prior to the first study dosing.
12. Pregnancy or breast-feeding.
13. Patients of reproductive age who are unable to use effective contraceptive measures in the period from the first dose of study drug to 180 days following the last dose of study drug. Female patients who have been amenorrheic for at least 12 months, have had a hysterectomy or oophorectomy, or have been surgically sterilized do not require contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: The incidence, nature, and severity of adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 in patients receiving the trial drug | up to 2 years
  Including grading of the incidence, nature, and severity of adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong